CLINICAL TRIAL: NCT07119450
Title: A Mass Balance Study of [14C] GZR18 in Chinese Overweight or Obese Male Subjects
Brief Title: The Study of [14C] GZR18
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZR18-BWM-105
Record Dates: First submitted 2025-07-09; First posted 2025-08-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Overweight; Obese; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GZR18 injection、[14C]GZR18 injection (Experimental)
  Interventions: Drug: GZR18 injection、[14C]GZR18 injection

INTERVENTIONS:
Drug: GZR18 injection、[14C]GZR18 injection — Participants will get a single dose of [14C]GZR18 injection

SUMMARY:
This trial is a Single-center, non-randomized, open-label, single-dose Mass Balance Study.

The study period of each subject consists of a screening period (D-21 to D-2), a baseline period (D-2 to D-1), a dosing and routine collection period (D1 to D36) and an intermittent collection and follow-up period (D36 to D78, during which subjects should visit the hospital once a week, 6 visits in total).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be fully informed, know and understand the content, process and possible treatment-related adverse events (TRAEs) before the study, and voluntarily sign a written informed consent form;
2. Chinese adult male subjects aged 18-55 (inclusive);
3. Body weight ≥ 50 kg;
4. Subjects with stable physical activity and lifestyle and relatively stable weight within 3 months prior to screening (as per inquiry);
5. Subjects have no sperm donation plan within 6 months after the last dose, and subjects and their partners have no pregnancy plan throughout the study and within 6 months after the last dose and voluntarily take effective contraceptive measures to avoid pregnancy of their partners.

Exclusion Criteria:

1. Subjects with other clinically significant diseases or medical history that may hinder the subject from following the study protocol and completing this study as judged by the investigator.
2. Subjects with abnormalities in vital signs, physical examination, routine laboratory tests (hematology, urinalysis, stool analysis + occult blood, blood chemistry and coagulation function), chest X-ray (AP view) or abdominal B-scan ultrasonography at screening or baseline, which are deemed clinically significant by the investigator; subjects with alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin exceeding the normal range at screening/baseline, which are deemed clinically significant by the investigator.
3. Subjects who suffer from dyspepsia, esophageal reflux, peptic ulcer or gallbladder disease within 3 months prior to dosing, or any gastrointestinal disease that may affect gastric emptying, or any surgical procedure (such as cholecystectomy, except for appendicitis surgery) that may affect drug metabolism or excretion; or plan to undergo surgery during the study.
4. Subjects who used any prescription drugs, OTC drugs, Chinese herbal medicines, food supplements (including vitamins, health food, etc.) within 14 days before dosing, or have other non-drug therapeutic factors affecting drug absorption, distribution, metabolism and excretion.
5. ubjects who have received any other investigational drug or participated in any other interventional clinical study within 3 months prior to screening, or still within 5 half-lives of a previously administered investigational drug at screening, whichever is longer.
6. Difficulty in blood collection or intolerance to venipuncture for blood collection.
7. Subjects who smoked > 5 cigarettes/day on average (or used an equivalent amount of nicotine products) in 6 months prior to screening, or are unwilling to abstain from tobacco products during the study.
8. Those who are not eligible for the study for other reasons as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | Through study completion, an average of 1 year
  The total radioactivity recovery at each interval and the cumulative total radioactivity recovery in excreta (urine and feces).
Primary Outcome Measure | Through study completion, an average of 1 year
  Percentage of parent drug and its metabolites (if applicable) in plasma in total radioactivity exposure in plasma; percentage of parent drug and its metabolites (if applicable) in urine and feces in administered dose; identification of major metabolites in plasma, urine, and feces.
Primary Outcome Measure | Through study completion, an average of 1 year
  Peak Plasma Concentration (Cmax)
Primary Outcome Measure | Through study completion, an average of 1 year
  Area under the plasma concentration versus time curve (AUC)
Primary Outcome Measure | Through study completion, an average of 1 year
  Ratio of total radioactivity concentration in whole blood to plasma
Primary Outcome Measure | Through study completion, an average of 1 year
  Time-To-Peak(Tmax)
Primary Outcome Measure | Through study completion, an average of 1 year
  Mean Residence Time
Primary Outcome Measure | Through study completion, an average of 1 year
  Half-Life Period（T1/2）

SECONDARY OUTCOMES:
PK parameters of GZR18 and its metabolites (if applicable) in plasma | Through study completion, an average of 1 year
  Peak Plasma Concentration (Cmax)
Safety Evaluation:Clinical safety evaluation during the study | Average of 1 year
  weight and height will be combined to report BMI in kg/m^2
PK parameters of GZR18 and its metabolites (if applicable) in plasma | Through study completion, an average of 1 year
  Area under the plasma concentration versus time curve (AUC)
PK parameters of GZR18 and its metabolites (if applicable) in plasma | through study completion, an average of 1 year
  Time-To-Peak(Tmax)
PK parameters of GZR18 and its metabolites (if applicable) in plasma | through study completion, an average of 1 year
  Mean Residence Time
PK parameters of GZR18 and its metabolites (if applicable) in plasma | through study completion, an average of 1 year
  Half-Life Period（T1/2）
Safety Evaluation:Clinical safety evaluation during the study | Average of 1 year
  laboratory tests (hematology, urinalysis, blood chemistry, coagulation function, stool analysis + occult blood and thyroid function)

CONTACTS AND LOCATIONS:
Locations (1):
- Study site 01, Beijing, China